CLINICAL TRIAL: NCT06060431
Title: Effectiveness of a Specific Pain Science Education Programme in Adolescent Students. Randomised Controlled Clinical Trial.
Brief Title: Effectiveness of a Pain Science Education Programme in Adolescent Students.
Acronym: EDEA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, Laura Menés Fernández, Principal Investigator, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 02/2022
Record Dates: First submitted 2023-09-18; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Chronic Pain; Pain; Pediatric ALL
MeSH Terms: conditions — Chronic Pain; Pain; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will carry out the sessions of the specific Pain Sciences program. This intervention is based on two educational sessions of 90 and 60 minutes each, separated by one week.
  Interventions: Other: Pain Science Education
- Control Group (No Intervention): The control group will not perform any specific intervention and will follow their usual academic curriculum.

INTERVENTIONS:
Other: Pain Science Education — The Pain Science Education program consists of two workshops, 90 and 60 minutes in length, one week apart. The content of the workshops aims to provide students with information about the contemporary pain paradigm and to re-conceptualize pain.
  Arms: Experimental group

SUMMARY:
The aim of this study is to analyze the effectiveness of a Pain Science Education program to improve the conceptualization of pain in adolescents between 11 and 13 years old, schooled in the first year of Compulsory Secondary Education.

DETAILED DESCRIPTION:
Design:

Randomized controlled clinical trial. The primary endpoint of the study was pain conceptualization recorded by a questionnaire.

Setting:

The participants were school-age children attending a different high school in the province of Barcelona.

Participants:

Of the 450 potential school participants, 306 agreed to participate. 13 pupils were excluded when applying the eligibility criteria, so the resulting sample was of 293

ELIGIBILITY:
Inclusion Criteria:

* to be schooled at the El Cim school
* to be between 10 and 16 years old (both included)
* to have or have had pain in the last month; to be able to read and write in Catalan and/or Spanish.

Exclusion Criteria:

* had an intellectual disability and/or cognitive impairment that interfered with their participation
* had not submitted the informed consent form duly completed and signed by their legal guardians

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 293 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Conceptualization of Pain Questionnaire (COPAQ) | 1 year
  The Conceptualization of Pain Questionnaire (COPAQ) consist of 15 items and asks respondents to respond if they believe the items/statements to be true or false, although they are allowed to respond undecided. A score of 0 is given to incorrect responses and those marked as undecided; the sum of all the correct answers gives the total score. The higher the score, the better the participant understands the concept of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Laura Menés Fernández, Vilanova i la Geltrú, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pate JW, Noblet T, Hush JM, Hancock MJ, Sandells R, Pounder M, Pacey V. Exploring the concept of pain of Australian children with and without pain: qualitative study. BMJ Open. 2019 Oct 28;9(10):e033199. doi: 10.1136/bmjopen-2019-033199. PMID 31662406
- [Background] Mankelow J, Ravindran D, Graham A, Suri S, Pate JW, Ryan CG, Martin D. An evaluation of a one-day pain science education event in a high school setting targeting pain related beliefs, knowledge, and behavioural intentions. Musculoskelet Sci Pract. 2023 Aug;66:102818. doi: 10.1016/j.msksp.2023.102818. Epub 2023 Jun 27. PMID 37418949
- [Background] Huguet A, Miro J. The severity of chronic pediatric pain: an epidemiological study. J Pain. 2008 Mar;9(3):226-36. doi: 10.1016/j.jpain.2007.10.015. Epub 2007 Dec 21. PMID 18088558